CLINICAL TRIAL: NCT01179763
Title: Analysis of Spectral Domain Optical Coherence Tomography Measurements in Amblyopia
Brief Title: Thickness of Retinal Layers in Amblyopia
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Se Yeul Oh, M.D., Samsung Medical Center
Other Study IDs: 2009-12-089
Record Dates: First submitted 2010-08-05; First posted 2010-08-11 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Amblyopia
Keywords: Amblyopia; Retinal layer thickness
MeSH Terms: conditions — Amblyopia | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Retinal layer thickness analysis: Optical coherence tomography will be conducted to analyze retinal layer thickness (safe examination)
  Interventions: Other: Optical coherence tomography

INTERVENTIONS:
Other: Optical coherence tomography — Spectral domain optical coherence tomography will be conducted once when patients are enrolled.
  Other Names: Spectralis Optical coherence tomography

SUMMARY:
The purpose of this study is to examine retinal layer thickness in amblyopia.

DETAILED DESCRIPTION:
Amblyopia is a visual disorder characterized by a reduction of vision that cannot be immediately improved by refractive correction or accounted for by clinically determined anatomic defects of the eye or visual pathway. Evidence for direct retinal changes in eyes with amblyopia has been controversial. It has been hypothesized that amblyopia may affect the postnatal maturation of the retina including the postnatal reduction of retinal ganglion cells. However, although some studies have found incrased retinal nerve fiber layer thickness in amblyopic eyes, others have found no significant differences. This sutdy will examine the retinal layer thickness in amblyopia and compare the retinal layer thickness between amblyopic eyes and nonamblyopic fellow eyes.

ELIGIBILITY:
Inclusion Criteria:

* Amblyopia

Exclusion Criteria:

* Other retinal disease
* Anisometropia
* Neurologic abnormalities

Ages: 4 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients in tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Retinal layer thickness | One month
  Optical coherence tomography scan will be conducted to analyze retinal layer thickness, when the patient are enrolled.

CONTACTS AND LOCATIONS:
Overall Officials: Sei Yeul Oh, M.D., Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Altintas O, Yuksel N, Ozkan B, Caglar Y. Thickness of the retinal nerve fiber layer, macular thickness, and macular volume in patients with strabismic amblyopia. J Pediatr Ophthalmol Strabismus. 2005 Jul-Aug;42(4):216-21. doi: 10.3928/01913913-20050701-03. PMID 16121551